CLINICAL TRIAL: NCT05774574
Title: Physiological and Appetitive Effects of Four Weeks of 60 mg/Day CBD Supplementation in an Adult Population
Brief Title: Physiological and Appetitive Effects of CBD Supplementation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Collaborators: Bridge Farm Nurseries Limited, Spalding, UK (Unknown)
Responsible Party: Principal Investigator, Lewis James, Senior Lecturer in Nutrition, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11031
Record Dates: First submitted 2023-01-16; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Appetitive Behavior; Adverse Effect; Metabolic Health
MeSH Terms: conditions — Appetitive Behavior | interventions — Cannabidiol; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD (Experimental): 1 mL hemp oil containing 60 mg/mL CBD, daily.
  Interventions: Dietary Supplement: Cannabidiol (CBD) supplementation
- Placebo (Placebo Comparator): 1 mL hemp oil containing 0 mg/mL CBD, daily.
  Interventions: Dietary Supplement: Placebo supplementation

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD) supplementation — Daily supplementation with 1 ml hemp oil containing 60 mg CBD, applied orally
  Arms: CBD
Dietary Supplement: Placebo supplementation — Daily supplementation with 1 ml hemp oil containing 0 mg CBD, applied orally
  Arms: Placebo

SUMMARY:
CBD may affect metabolic control and energy intake. However, there is currently little data regarding these specific outcomes in humans. Therefore, this study will investigate whether four weeks of supplementation with 60 mg/day CBD affects energy intake at a single meal, and or fasting blood-based markers of appetite regulation and metabolic health. Healthy, adult volunteers will be assigned to placebo or CBD supplementation, in a randomized controlled trial, comparing changes in outcomes across the supplementation period between groups.

ELIGIBILITY:
Exclusion Criteria:

* No history of any substance abuse
* Have used tobacco regularly (>2x in a week) within the past 6 months
* Are suffering from any condition that may affect study outcomes
* Currently use any prescription or over-the-counter medications (except for hormonal contraception and simple painkillers)
* Have given a standard blood donation within 30 days of screening
* Are currently pregnant or lactating
* Are allergic/intolerant to any ingredients in food items we provide during the study (relevant allergens: oats, milk)

Inclusion Criteria:

* Males and females, aged 18-50, who do not meet the exclusion criteria

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-05 (Estimated)

PRIMARY OUTCOMES:
Energy Intake | Baseline and after 4 weeks supplementation
  Self-selected energy intake at an ad libitum mixed meal

SECONDARY OUTCOMES:
CBD | Baseline and after 4 weeks supplementation
  CBD circulating in plasma
Liver transaminases | Baseline and after 4 weeks supplementation
  AST and ALT circulating in plasma
Hormones implicated in appetite regulation | Baseline and after 4 weeks supplementation
  Hormones implicated in appetite regulation (e.g., leptin and ghrelin) circulating in plasma
Lipoproteins | Baseline and after 4 weeks supplementation
  Lipoproteins (e.g., total cholesterol, HDL-C and LDL-C) circulating in plasma
Glucose | Baseline and after 4 weeks supplementation
  Glucose circulating in plasma
Triglycerides | Baseline and after 4 weeks supplementation
  Triglycerides circulating in plasma
Insulin | Baseline and after 4 weeks supplementation
  Insulin circulating in plasma
Subjective appetite (hunger, fullness, desire to eat) | Baseline and after 4 weeks supplementation
  Measured using pen and paper scales (scored 'not at all' [0 mm] to 'extremely' [100 mm])
self-reported adverse events | During 4 weeks supplementation
  Adverse events reported in diary by participants

CONTACTS AND LOCATIONS:
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual data for study outcomes will be shared on the Loughborough University Research Repository
Time Frame: Permanently, after publication of study findings.